CLINICAL TRIAL: NCT04440670
Title: Effect of Autologous Cord Blood Mononuclear Cells for Prevention of Bronchopulmonary Dysplasia or Death in Extremely Preterm Neonates: a Placebo-controlled Randomized Multicenter Trial
Brief Title: Effect of Autologous Cord Blood Mononuclear Cells for Prevention of Bronchopulmonary Dysplasia or Death in Extremely Preterm Neonates
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Collaborators: Foshan Fuxing Chancheng Central Hospital (Unknown); Foshan Women's and Children's Hospital (Other); Hexian Memorial Affiliated Hospital of Southern Medical University (Unknown); Heyuan Women and Children Hospital (Unknown); Dongguan Women and Children Hospital (Unknown); Guangzhou Huadu Women and Children Hospital (Unknown); Shunde Women and Children Hospital (Unknown); Guangdong Cord Blood Bank (Industry); Huangdu Distric Women and Children Hospital (Unknown); Longgang Distric Women and Children Hospital,Shenzhen (Unknown); BoAi Hospital of Zhongshan (Other); Huizhou first Women and Children Hospital (Unknown); Huizhou second Women and Children Hospital (Unknown)
Responsible Party: Principal Investigator, yang jie, Professor, Guangdong Women and Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Guang dong W C H
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: BPD
Keywords: Autologous cord blood mononuclear cells; bronchopulmonary dysplasia; extremely preterm neonates
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: In this prospective, randomized controlled double-blind multi-center clinical trial, 140 preterm neonates less than 28 weeks are randomly assigned to receive intravenous autologous cord blood mononuclear cells infusion (5×107cells/kg) or placebo ( normal saline) within 24 hours after birth in a 1:1 ratio using a central randomization system.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A hospital ethics committee reviewed the study data during the trials. None of them were involved in the study or aware of the treatment-group assignments of the infants. Only nurses and physicians staff conducted the infusion were aware of the treatment assignment, and these individuals had no contact with the staff who collected and analyzed the patients data. The parents are not aware of the assignment. This study is double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACBMNC infusion group (Experimental): Those assigned to the ACBMNC group will receive intravenous autologous cord blood mononuclear cells infusion within 24 h after birth. Cell dose for all patients was targeted at 5×107 cells per kilogram.
  Interventions: Biological: autologous cord blood mononuclear cells
- control group (Placebo Comparator): Those in control group will receive an infusion of a placebo solution which is normal saline with the same volume.
  Interventions: Biological: normal saline

INTERVENTIONS:
Biological: autologous cord blood mononuclear cells — preterm neonates less than 28 weeks are assigned to receive intravenous autologous cord blood mononuclear cells infusion (5×107cells/kg) within 24 hours after birth
  Arms: ACBMNC infusion group
Biological: normal saline — preterm neonates less than 28 weeks are assigned to receive normal saline within 24 hours after birth
  Arms: control group

SUMMARY:
This is the first and largest randomized, controlled, blinded trial that evaluates the efficacy of autologous cord blood mononuclear cells infusion as a prevention therapy for BPD or death. The results of this trial will provide valuable clinical evidence for recommendations on the management of BPD in extremely preterm infants. In this prospective, randomized controlled double-blind multi-center clinical trial, 140 extremely preterm neonates less than 28 weeks are randomly assigned to receive intravenous autologous cord blood mononuclear cells infusion (targeted dose of 5×107cells/kg but no less than 1×107cells/kg) or placebo ( normal saline) within 24 hours after birth in a 1:1 ratio using a central randomization system. The primary outcome is survival without bronchopulmonary dysplasia at 36 weeks of postmenstrual age or discharge home. The secondary outcomes will include mortality rate, BPD severity, other common preterm complication rate, respiratory support duration, the length and cost of hospitalization and long term outcomes after two years follow up post infusion.

DETAILED DESCRIPTION:
Study design and settings:

This present study will be a randomized, placebo-controlled, double-blinded, multi-center trial to be conducted at 12 medical centers in tertiary hospitals with Neonatal Intensive Care Unit that were selected by the expert committee. A total of 140 neonates fulfilling the eligibility criteria will be enrolled. Subsequently, the participants will be randomly divided into two groups (ACBMNC infusion group and control (placebo) group ) in a ratio of 1:1.

Sample size:

Based on our previous study and others' study, we found the ACBMNC infusion was effective in reducing respiratory support duration in preterm infants. The rate of BPD among extremely preterm infants in our NICU was 60% (pA). What we expect to be an intended (or at least acceptable) effect of the ACBMNC infusion is 25 % reduction in frequency of BPD(pB:35%). To detect this difference with a sensitivity of 80% and an error probability of 5%, at least 59 patients per randomization group will be required using the following formula:

n=(pA(1-pA)/κ+pB(1-pB))((z1-α/2+z1-β)/(pA-pB))2 To account for the possibility of as high as 20% loss to follow-up, our estimated sample size is 140 cases totally.

Objectives:

Primary objective： The primary objective of this trial is to evaluate the efficacy of ACBMNC infusion in preventing bronchopulmonary dysplasia or death at 36 weeks of postmenstrual age or discharge home in extremely preterm infants.

Secondary objectives：

* To compare the mortality rate at 36 weeks of postmenstrual age.
* To compare the BPD severity
* To compare the rate of other common preterm complications included intraventricular hemorrhage (IVH), necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), respiratory distress syndrome (RDS), ventilation-associated pneumonia (VAP), hypoxic ischemic encephalopathy (HIE), late onset sepsis (LOS) and anemia.To compare the duration of mechanical ventilation and oxygen therapy in two groups
* To determine re-intubation rate and time return to BW
* To compare the duration of antibiotic usage
* To determine the long term outcomes after two years follow up

Participants:

Inclusion criteria:

Infants fulfilling all the following inclusion criteria will be enrolled in this trial: 1. born at study hospital; 2. singleton birth; 3. less than 28 weeks GA 4.Signed informed consent obtained; 5. had available umbilical cord blood (UCB).

Exclusion criteria:

Those infants are excluded if they were 1. with severe congenital abnormalities; 2.with maternal clinical chorioamnionitis 3. the mother was positive for hepatitis B (HBsAg and/or HBeAg) or C virus (anti-HCV), syphilis, HIV (anti-HIV-1 and -2) or IgM against cytomegalovirus, rubella, toxoplasma and herpes simplex virus.

Trial treatment methods:

Soon after the preterm infant was deliveried, written consent was signed by the parents, and autologous cord blood infusion was applied to the baby in addition to routine pulmonary surfactant replacement, and mechanical ventilation support as indicated. Those assigned to the ACBMNC group received an infusion of ACBMNC with 24 h after birth. Those in control group received an infusion of a placebo solution which is normal saline with the same volume. Cell dose for all patients was targeted at 5×107 cells per kilogram.

ELIGIBILITY:
Inclusion Criteria:

Infants fulfilling all the following inclusion criteria will be enrolled in this trial: 1. born at study hospital; 2. singleton birth; 3. less than 28 weeks GA 4.Signed informed consent obtained; 5. had available umbilical cord blood (UCB).

Exclusion Criteria:

Those infants are excluded if they were 1. with severe congenital abnormalities; 2.with maternal clinical chorioamnionitis 3. the mother was positive for hepatitis B (HBsAg and/or HBeAg) or C virus (anti-HCV), syphilis, HIV (anti-HIV-1 and -2) or IgM against cytomegalovirus, rubella, toxoplasma and herpes simplex virus.

Ages: 0 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
frequency of bronchopulmonary dysplasia or death | 36 weeks of postmenstrual age or discharge home whichever comes first.
  The frequency of bronchopulmonary dysplasia or death at 36 weeks of postmenstrual age or discharge home whichever comes first.

SECONDARY OUTCOMES:
mortality | 36 weeks of postmenstrual age or the discharge
  The mortality rate.
  * Incidence of other preterm complications including intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), respiratory distress syndrome (RDS), ventilation-associated pneumonia (VAP), late onset sepsis (LOS) and anemia .
  * Duration of hospitalization.
  * Duration of mechanical ventilation and oxygen therapy
  * The frequency of re-intubation.
  * The time (days) return to BW.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, Study Chair — Guangdong Women and Children Hospital
Locations (2):
- China (2):
  - Ren Xuejun, Dongguan, Guangdong
  - Jie Yang, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Yes
public
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: all time
Access Criteria: all